CLINICAL TRIAL: NCT00218413
Title: A Phase 2 Study to Assess Safety and Immunogenicity of Five Doses of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX) Administered to Smokers
Brief Title: Safety and Effectiveness of NicVAX in Treating Nicotine Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Arjen DeVos/ Senior Director, Medical Affairs and Clinical Research, Nabi Biopharmaceuticals
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-17894-2; Nabi-4505; R01-17894-2; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-11

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
Keywords: Vaccine; Immunogenicity; Randomized Controlled Trial; Addiction
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Behavior, Addictive | interventions — NicVAX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Biological: NicVAX
- 2 (Experimental)
  Interventions: Biological: NicVAX
- 3 (Experimental)
  Interventions: Biological: NicVAX
- 4 (Experimental)
  Interventions: Biological: NicVAX
- 5 (Experimental)
  Interventions: Biological: NicVAX

INTERVENTIONS:
Biological: NicVAX — 100 μg, Formulation A, on Days 0, 21, 42, 91 & 182
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 1
Biological: NicVAX — 200 μg, Formulation A, on Days 0, 21, 42, 91 & 182
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 2
Biological: NicVAX — 200 μg, Formulation B, on Days 0, 21, 42m 91 & 182
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 3
Biological: NicVAX — 300 μg, Formulation B, on Days 0, 21, 42, 91 & 182
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 4
Biological: NicVAX — 400 μg, Formulation B, on Days 0, 21, 42, 91 & 182
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 5

SUMMARY:
Nicotine is highly addictive and many individuals are unable to quit smoking even with treatment. The purpose of this study is to determine the effectiveness of various doses of NicVAX in treating nicotine dependent individuals.

DETAILED DESCRIPTION:
Tobacco use is the single leading preventable cause of death in the United States. Nicotine is an alkaloid that is derived from the tobacco plant responsible for the psychoactive and addictive effects of smoking. Immunotherapy may be useful in preventing and treating nicotine dependent individuals. NicVAX is a nicotine vaccine, a type of immunotherapy that may be effective in smoking cessation and preventing relapse to nicotine. The purpose of this study is to evaluate the safety and efficacy of various dosing levels and dosing frequencies of NicVAX in treating nicotine dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker
* Good general health, including mental health
* Alveolar carbon monoxide level greater than or equal to 10 ppm

Exclusion Criteria:

* Prior exposure to NicVAX
* Known allergy to any of the components of NicVAX
* Use of any smoking cessation aide
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Anti-nicotine Antibody concentrations | 19 time points from Day 0 to 365

SECONDARY OUTCOMES:
Smoking cessation | periods of 2 weeks, 4 weeks, or 12 weeks duration
Fagerstrom Test for Nicotine Dependence | 7 time points from Day 0 to 365
Safety: vaccine reactogenicity | 7 days after each dose
Safety: adverse events | Day 0-365

CONTACTS AND LOCATIONS:
Overall Officials: Gary Horwith, Principal Investigator — Nabi Biopharmaceuticals; Arjen De Vos, MD, PhD, Principal Investigator — Nabi Biopharmaceuticals
Locations (1):
- University of Maastricht, Maastricht, Netherlands